CLINICAL TRIAL: NCT01990885
Title: A Two-Part, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Systemic Exposure of Single Escalating Administrations and Repeated Administration of BL-7010 in Well-Controlled Celiac Patients
Brief Title: Safety and Systemic Exposure Study of BL-7010 in Well-Controlled Celiac Patients.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioLineRx, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BL-7010.01
Record Dates: First submitted 2013-11-17; First posted 2013-11-25 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: A Two-Part, Randomized, Double-Blind, Placebo-Controlled Study To Evaluate The Safety And Systemic Exposure Of Single Escalating Administrations And Repeated Administration Of Bl-7010 In Well-Controlled Celiac Patients
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- Cohort A (Experimental): Each subject will receive a single administration of either BL-7010 (at different amounts) or matching Placebo on 3 treatment occasions in a randomized double-blind fashion
  Interventions: Drug: BL-7010; Drug: Placebo
- Cohort B (Experimental): Each subject will receive a single administration of either BL-7010 (at different amounts) or matching Placebo on 3 treatment occasions in a randomized double-blind fashion
  Interventions: Drug: BL-7010; Drug: Placebo
- Cohort C (Experimental): Each Subject will receive either BL-7010 or Placebo 3 times a day for 14 days(amount to be based on results from Cohorts A and B) in a randomized double-blind fashion
  Interventions: Drug: BL-7010; Drug: Placebo
- Cohort D (Experimental): Each Subject will receive either BL-7010 or Placebo 3 times a day for 14 days(amount to be based on results from previous cohorts) in a randomized double-blind fashion
  Interventions: Drug: BL-7010; Drug: Placebo
- Cohort E (Experimental): Each Subject will receive either BL-7010 or Placebo 3 times a day for 14 days(amount to be based on results from previous cohorts) in a randomized double-blind fashion
  Interventions: Drug: BL-7010; Drug: Placebo

INTERVENTIONS:
Drug: BL-7010
  Other Names: BL7010
Drug: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety of different amounts of BL-7010 in single oral administration and in repeated oral administration to well-controlled celiac patients. Another purpose is to evaluate if BL-7010 is absorbed by the body or not.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18-75 years who have signed an informed consent form
* Body mass index (BMI) between 18.5-29.9, inclusive
* Documented history of biopsy-proven celiac disease.
* Adherence to a gluten-free diet for the last 6 months prior to randomization
* TG2 and EMA antibody (IgA) negative
* Women of childbearing potential and all men must agree to use an approved form of contraception
* Ability and willingness to understand and comply with study procedures and to give written informed consent prior to enrollment.

Exclusion Criteria:

* IgA deficiency.
* History of IgE-mediated reactions to gluten.
* Other food sensitivities or allergies.
* Use of oral steroids, biologics, immunosuppressants or non-steroidal anti-inflammatory drugs 6 months prior to entry (screening).
* Female subjects who are pregnant or breastfeeding.
* Clinically significant, concomitant gastrointestinal disease.
* Have clinically significant current or historical medical problems such as diabetes mellitus, clinically significant cardiac arrhythmias, arteriosclerotic heart disease, renal insufficiency or failure, autoimmune disease, history of malignant melanoma or history of cancer (excluding basal cell carcinoma) within the past 5 years prior to screening.
* Subjects receiving drugs or oral devices that, in the opinion of the Investigator, possible ineffective treatment with these drugs/oral devices for a duration of two weeks will put the subject at a medical risk
* Uncontrolled complications of celiac disease.
* Any other condition that in the opinion of the Investigator will place the subject at risk or prevent protocol compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | For Part 1 subjects will be followed for up to 7 weeks from time of first administration. For Part 2 subjects will be followed for up to 4 weeks from time of first administration
Significant change from baseline in vital signs and 12-lead ECG parameters | For Part 1 subjects will be followed for up to 7 weeks from time of first administration. For Part 2 subjects will be followed for up to 4 weeks from time of first administration
Significant change from baseline in laboratory safety parameters | For Part 1 subjects will be followed for up to 7 weeks from time of first administration. For Part 2 subjects will be followed for up to 4 weeks from time of first administration

SECONDARY OUTCOMES:
Plasma levels of BL-7010 | Over a 24 hour period

CONTACTS AND LOCATIONS:
Overall Officials: Markku Mäki, Professor, Principal Investigator — Tampere University
Locations (2):
- Finland (2):
  - FinnMedi Clinical Trial Center, Tampere
  - CRST Clinical Research Services, Turku